CLINICAL TRIAL: NCT07086937
Title: To Compare the Efficacy of Nitrazoxinide Based Triple Therapy Versus Standard Triple Therapy for Eradication of Helicobacter Pylori Infection in Children at a Tertiary Care Hospital
Brief Title: Efficacy of Nitazoxanide Based Therapy vs Standard Triple Therapy in H-pylori in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dr-Shumaila-ZUH
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — nitazoxanide; Metronidazole; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NTZ-based group (Experimental): Children in NTZ-based group were given triple regimen, i.e., nitazoxanide, PPI, and clarithromycin for 14 days.
  Interventions: Drug: Nitazoxanide; Drug: PPI; Drug: Clarithromycin
- MTZ-based group (Experimental): Children in MTZ-based triple regimen received metronidazole, PPI, and clarithromycin for 14 days.
  Interventions: Drug: Metronidazole; Drug: PPI; Drug: Clarithromycin

INTERVENTIONS:
Drug: Nitazoxanide — Children were given nitazoxanide, PPI, and clarithromycin for 14 days.
  Arms: NTZ-based group
Drug: Metronidazole — Children received MTZ, PPI, and clarithromycin for 14 days.
  Arms: MTZ-based group
Drug: PPI — Children were given omeprazole for 14 days.
Drug: Clarithromycin — Children were given clarithromycin for 14 days.

SUMMARY:
This study aimed at comparing the efficacy of nitazoxanide-based triple therapy versus standard triple therapy for eradication of Helicobacter pylori infection in children at a tertiary care hospital.

DETAILED DESCRIPTION:
The findings could guide clinical practice and influence guidelines, improving the management of H. pylori infections in the pediatric population. Not much local data also exists comparing the effectiveness of adding nitazoxanide to the standard triple therapy in children with H. pylori infection. If nitazoxanide-based therapy proves superior, it could reduce the incidence of antibiotic resistance associated with standard triple therapy.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* Aged 2 to 12 years
* With symptoms like abdominal pain, nausea, vomiting, or other related gastrointestinal symptoms
* Diagnosed with H. pylori based on urea breath test

Exclusion Criteria:

* Liver cirrhosis
* Renal impairment
* Previous gastric or duodenal surgery or malignancy
* History of receiving H. pylori treatment
* Past 6 weeks history of using antacids, H2 receptor antagonists, anticoagulants, or antibiotics

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy | 6 weeks
  The patients were considered clinically cured if they had a negative H. pylori stool Ag test and were free of symptoms at 6 weeks after starting treatment, or otherwise failure was labeled.

CONTACTS AND LOCATIONS:
Overall Officials: Shumaila Waseem, Principal Investigator — Ziauddin University Karachi; Heena Raees, FCPS, Study Director — Ziauddin University Karachi
Locations (1):
- Ziauddin University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.